CLINICAL TRIAL: NCT03760367
Title: Investigation of the Instant Tooth Whitening Effect of a Silica Toothpaste Containing Blue Covarine - a Randomized Controlled Clinical Trial
Brief Title: Investigation of the Instant Tooth Whitening Effect of a Silica Toothpaste Containing Blue Covarine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IOOS_TA_01_2018
Record Dates: First submitted 2018-11-19; First posted 2018-11-30 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2018-11

CONDITIONS: Tooth Whitening
Keywords: blue covarine; numeric analogue scale; spectrophotometry; tooth bleaching

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups - blue covarine toothpaste and control toothpaste group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are randomly assigned to one of the two arms and perform the treatment without knowing whether they use the blue covarine toothpaste or the control toothpaste. Treatment outcomes are assessed by a) a blinded operator and b) the blinded participants in a different room. Allocation of treatment groups will be revealed to the principal investigator after all data have been collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue Covarine Toothpaste (Experimental): After a short video introduction to the bass technique, participants brush their teeth once with a silica toothpaste containing blue covarine (Pepsodent White Now Gold, 1 g) for 2 min, starting with the upper front teeth. Thereafter, participants rinse their mouth with of tap water.
  Interventions: Other: Blue covarine toothpaste
- Control Toothpaste (Active Comparator): After a short video introduction to the bass technique, participants brush their teeth once with a silica toothpaste (Colgate Advanced Whitening, 1 g) for 2 min, starting with the upper front teeth. Thereafter, participants rinse their mouth with of tap water.
  Interventions: Other: Control toothpaste

INTERVENTIONS:
Other: Blue covarine toothpaste — 2 min toothbrushing with 1 g of Pepsodent White Now Gold
  Other Names: Pepsodent White Now Gold
  Arms: Blue Covarine Toothpaste
Other: Control toothpaste — 2 min toothbrushing with 1 g of Colgate Advanced Whitening
  Other Names: Colgate Advanced Whitening
  Arms: Control Toothpaste

SUMMARY:
The study investigates the effect of toothbrushing with a toothpaste containing blue covarine compared to a control toothpaste without blue covarine on tooth color. Participants brush their teeth once with either the blue covarine containing toothpaste or a control toothpaste for two minutes. Before and after brushing, tooth color is assessed with a spectrophotometer. Moreover, satisfaction of the participants with their tooth color is assessed using a numeric analogue scale before and after treatment.

The null hypotheses are that neither brushing with the toothpaste containing blue covarine nor brushing with the control toothpaste change a) the tooth color and b) the satisfaction of the participants with their tooth color.

DETAILED DESCRIPTION:
Participants are recruited by advertizing in several public areas in Aarhus, Denmark.

Written and oral information on the study is provided, eligibility criteria are checked, and informed consent is given by the participants.

The upper front teeth of the participants are cleaned with pumice and a rubber cup by operator A.

Participants look at the color of their upper front teeth with a mirror, in a room with controlled lighting conditions.

Thereafter, participants rate their satisfaction with the color of their teeth using an 11-point aesthetic numeric analogue scale.

Tooth color is assessed by operator B using a spectrophotometer (VITA Easyshade Advance) and a positioning device to standardize measurements. Measurements are performed in a room with controlled lighting conditions. VITA SYSTEM 3D-MASTER color, L*, a* and b* are recorded.

Participants are then randomly assigned to either the blue covarine toothpaste group or the control toothpaste group.

They are given a short video introduction to the Bass toothbrushing technique by operator C (caregiver).

Operator C provides a toothbrush and 1 g of either blue covarine toothpaste or control toothpaste, according to the randomization scheme.

Participants brush their teeth for two min, starting with the upper front teeth, and then rinse their mouth with tap water.

Thereafter, participants look again at the color of their upper front teeth with a mirror, in the same room as before treatment.

They rate their satisfaction with the color of their teeth using the 11-point aesthetic numeric analogue scale.

Moreover, they rate the color difference before and after treatment on an 11-point aesthetic numeric analogue scale.

Again, tooth color is assessed by operator B using a spectrophotometer (VITA Easyshade Advance) and a positioning device to standardize measurements. Measurements are performed in the room with controlled lighting conditions. Again VITA SYSTEM 3D-MASTER color, L*, a* and b* are recorded.

The null hypotheses of the study are that neither brushing with the toothpaste containing blue covarine nor brushing with the control toothpaste change a) the tooth color and b) the satisfaction of the participants with their tooth color.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Dental caries in the upper front teeth
* Intrinsic stain of the upper front teeth, including tetracyclin stains, fluorosis, and staining due to pulpitis or pulp necrosis
* Dental restorations in the upper front teeth, including fillings, veneers, crowns, and root canal fillings
* Dental anomalies of the upper front teeth, including molar incisor hypomineralisation, amelogenesis imperfecta, and dentinogenesis imperfecta

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
3D VITA SYSTEM 3D-MASTER tooth color change | Tooth color is measured twice, right before (baseline) and immediately after toothbrushing.
  Tooth color change of the upper right first incisor is assessed after toothbrushing compared to baseline using a spectrophotometer.
Change of participant satisfaction with the tooth color | Participant satisfaction is assessed twice, right before (baseline) and immediately after toothbrushing.
  Change of participant satisfaction with the color of their upper front teeth is assessed after toothbrushing compared to baseline using an 11 step aesthetic numeric analogue scale (ANA scale, Funk et al., 2011; DOI: https://doi.org/10.1016/j.jcms.2011.07.018).

SECONDARY OUTCOMES:
Change of blue-yellow color component of the tooth (b* in the CIELAB color space) | The blue-yellow color component is assessed twice, right before (baseline) and immediately after toothbrushing.
  The change of the blue-yellow color component of the upper right first incisor is assessed after toothbrushing compared to baseline using a spectrophotometer.
Change of the green-red color component of the tooth (a* in the CIELAB color space) | The green-red color component is assessed twice, right before (baseline) and immediately after toothbrushing.
  The change of the green-red color component of the upper right first incisor is assessed after toothbrushing compared to baseline using a spectrophotometer.
Change of the tooth lightness value (L* in the CIELAB color space) | The tooth lightness is assessed twice, right before (baseline) and immediately after toothbrushing.
  The change of lightness of the upper right first incisor is assessed after toothbrushing compared to baseline using a spectrophotometer.
Participant evaluation of tooth color change | The color change of the upper front teeth is assessed once: immediately after toothbrushing.
  The color change of their upper front teeth is assessed visually by the participants using an 11 step aesthetic numeric analogue scale (ANA scale, Funk et al., 2011; DOI: https://doi.org/10.1016/j.jcms.2011.07.018).

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schlafer, Dr., Principal Investigator — Aarhus University, Department of Dentistry and Oral Health
Locations (1):
- Aarhus University, Department of Dentistry and Oral Health, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to general data protection regulations, individual participant data will not be made available publicly. Summary data will be made available upon publication of the results.